CLINICAL TRIAL: NCT01240824
Title: A Phase I Trial to Determine the Safety, Tolerability and Maximum Tolerated Intravesical Dose of Aminophylline With BCG in Patients With Non-invasive Bladder Cancer
Brief Title: Study of BCG + Aminophylline Toxicity When Used in the Treatment of Bladder Cancer
Acronym: BCG
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 14585
Record Dates: First submitted 2010-11-11; First posted 2010-11-15 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; urothelial carcinoma; transitional cell carcinoma bladder; ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Aminophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BCG + aminophylline (Experimental): Bacillus Calmette-Guerin (BCG) plus one of three escalating doses of aminophylline administered intravesically.
  Interventions: Drug: aminophylline

INTERVENTIONS:
Drug: aminophylline — One of three escalating doses of aminophylline (3 mg/kg, 6 mg/kg and 9 mg/kg) administered intravesically

SUMMARY:
The purpose of this study is to evaluate whether a new potential treatment for non invasive bladder cancer is safe and if it leads to side effects such as irregular heart rate, agitation, or burning with urination. Patients who have early stage bladder cancer and will be receiving BCG, a bladder cancer therapy as recommended by a doctor, will be asked to participate in a study where they are given the standard BCG followed by the experimental drug, aminophylline. Although we hope this medicine may one day prove to help bladder cancer patients, at the current time we do not know if it has any benefits at all. We have data in mice that suggest that aminophylline slows the growth of tumors when coupled with BCG.

DETAILED DESCRIPTION:
Before using the combination of BCG and aminophylline clinically, we need to first determine if aminophylline is safe, when placed directly into the bladder of patients who have bladder cancer. We will give it along with BCG (Bacillus Calmette-Guerin) - a medication put into the bladder through a catheter tube to treat bladder cancer.

We also would like to determine the maximum dose of aminophylline that can be safely given and how the drug is absorbed and used by the body as well as document side effects when aminophylline is given in the bladder.

This is a study about aminophylline instilled into the bladder. Aminophylline has not been proven to be safe or a helpful treatment for bladder cancer. It is considered an experimental drug as used in this protocol for bladder cancer. Aminophylline has not been given to anyone who has bladder cancer. Aminophylline is approved by the U.S. Food and Drug Administration (FDA ) to give directly into the bloodstream for the treatment of asthma. We intend to use it at doses much lower than that used for asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 40 years of age because in patients younger than that the natural history is different.
2. Histologically proven bladder cancer that is NOT muscle invasive (Ta or T1)
3. Transurethral resection of Bladder Tumor (TURBT) at least 2 weeks prior to first instillation
4. ECOG performance status of 0 or 1.
5. Informed consent obtained from patient before enrollment.
6. English is primary language
7. Patients undergoing initial 6 week BCG therapy (BCG naïve)
8. Patients undergoing 3 week BCG maintenance therapy.

Exclusion Criteria:

1. Hypersensitivity reaction or contraindication to aminophylline or theophylline
2. Pregnancy (confirmed by a serum human chorionic gonadotropin pregnancy test) or breast feeding).
3. Hepatic insufficiency as defined by an abnormal AST or ALT.
4. Known arrhythmias or heart failure as defined by class II or greater cardiovascular disease according to the New York Heart Associations functional criteria
5. Immunocompromised
6. Seizure disorder.
7. Current treatment with oral theophylline or any other methylxanthine derivative.
8. Active urinary tract infection by nitrite positive urine dip or gross hematuria
9. Reduced dosing of BCG or BCG failures who have experienced bladder cancer recurrrence.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity | Week 6
  Any cardiac arrythmia or seizure activity, > grade 2 allergic reactions, fever 101.5 for > 48 hours, > grade 1 insomnia, > grade 1 involuntary movements, > grade 2 nausea / vomiting, > grade 2 bladder spasms, dysuria or pelvic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy L Krupski, M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Urology Department, Charlottesville, Virginia, United States